CLINICAL TRIAL: NCT04699175
Title: A Phase Ⅱ, Multicenter, Randomized, Single-Blind, Placebo-Controlled, Evaluation of the Safety, Efficacy of HR021618 for Pain Management Following Orthopaedic Surgery
Brief Title: A Trial of HR021618 in Postsurgical Pain Management
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR021618-202
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2020-12

CONDITIONS: Postsurgical Pain Management

STUDY DESIGN:
Intervention Model Description: HR021618 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental)
  Interventions: Drug: HR021618
- Treatment group B (Experimental)
  Interventions: Drug: HR021618
- Treatment group C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HR021618 — Treatment group A:HR021618; high dose
  Arms: Treatment group A
Drug: HR021618 — Treatment group B:HR021618; low dose
  Arms: Treatment group B
Drug: Placebo — Treatment group C: HR021618 blank preparation.
  Arms: Treatment group C

SUMMARY:
The study is being conducted to evaluate the efficacy, safety of HR021618 and to explore the reasonable dosage of HR021618 for Pain Management after Orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective Orthopaedic surgery
3. Male or female
4. Meet the weight standard
5. Conform to the ASA Physical Status Classification Postoperative randomization criteria Exclusion Criteria

1、 Sufficient pain to require IVanalgesia assessed by NRS ranging 2、 No evidence of organ insufficiency, or any other abnormality, during or following surgery

Exclusion Criteria:

1. History of major surgery
2. History of active or high-risk bleeding disorders
3. History of myocardial infarction or coronary artery bypass
4. History or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study
5. Abnormal values in the laboratory
6. Have a known allergy to meloxicam or any excipient of HR021618, , aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs) or to any peri- or postoperative medications used in this study
7. Use other drugs that affect the analgesic effect before randomization, and the time from the last use to randomization is shorter than 5 half-lives
8. Planned/actual admission to the intensive care unit
9. Pregnant or nursing women
10. No birth control during the specified period of time
11. Participated in clinical trials of other drugs (received experimental drugs)
12. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-08 (Estimated)

PRIMARY OUTCOMES:
Usage of Morphine, Post Surgery | 0 hour to 24 hours after IP administration
  Change in the amount of morphine use (in milligrams) by subjects in each treatment group for a 24 hour period post IP administration.

SECONDARY OUTCOMES:
Usage of Morphine, Post Surgery at other intervals | 0 hour to 48 hours after IP administration
  Change in the amount of morphine use (in milligrams) by subjects in each treatment group for 0-48 hours after IP administration.
Pain intensity assessed using an 11-point NRS ranging | Baseline till 48 hours post IP administration
  11-point NPRS ranging from a score of 0 to 10.
Pain relief assessed using an 5-point likert scale | Baseline till 48 hours post IP administration
  5-point likert scale from a score of 0 to 4.
Time to First Dose of Rescue Analgesia | 0 hour to 48 hours after IP administration
  Time to first rescue was calculated as the elapsed time from administration of Dose 1 to the administration of the first dose of rescue analgesia.
Frequency of Doses of Rescue Analgesia Utilized Per Subject | 0 hour to 48 hours after IP administration
  Rescue analgesia was available to subjects with inadequately controlled pain upon request.
Proportion of subjects who received Rescue Analgesia | 0 hour to 48 hours after IP administration
  Proportion of rescue was calculated as the elapsed time from administration of Dose 1 to the administration of the first dose of rescue analgesia.
Patient Global Assessment (PGA) of Pain Control | 0 hour to 48 hours after IP administration
  PGA of pain control was evaluated by subject reported degree of pain control according to a 5 point scale (0-4)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China